CLINICAL TRIAL: NCT02214667
Title: Treating Co-Occurring Substance Use and Mental Disorders Among Jail Inmates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit enough participants
Sponsor: RTI International (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34DA036791 (NIH)
Record Dates: First submitted 2014-08-10; First posted 2014-08-12 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Co-occurring Mental and Substance Use Disorders; Crime; Criminogenic Thinking; Implementation; Adaptation
Keywords: Jail; co-occurring disorders; implementation; acceptability; feasibility; fidelity
MeSH Terms: conditions — Substance-Related Disorders | interventions — Jails

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DDMI-IGT (Experimental): Subjects randomized to the experimental condition will receive adapted versions of dual-diagnosis motivational interviewing ([DDMI] one session before release from jail) and integrated group therapy ([IGT] 12 community-based sessions over a 2-month period).
  Interventions: Behavioral: Dual-diagnosis motivational interviewing (DDMI); Behavioral: Integrated group therapy (IGT)
- Usual care (Active Comparator): Subjects randomized to the usual care condition will receive jail and community-based behavioral health services.
  Interventions: Behavioral: Jail and community-based behavioral health services

INTERVENTIONS:
Behavioral: Dual-diagnosis motivational interviewing (DDMI) — DDMI is an evidence-based adaptation to motivational interviewing. DDMI incorporates an integrated framework and accommodates cognitive impairments and disordered thinking associated with co-occurring substance use and mental disorders.
  Arms: DDMI-IGT
Behavioral: Integrated group therapy (IGT) — IGT is an evidence-based practice for treating co-occurring disorders. IGT focuses on relapse prevention by reducing substance use and stabilizing psychiatric symptoms.
  Arms: DDMI-IGT
Behavioral: Jail and community-based behavioral health services — Existing behavioral health service programs
  Arms: Usual care

SUMMARY:
Treatment adaptation and implementation study for adult jail inmates with co-occurring substance use disorders.

DETAILED DESCRIPTION:
We will adapt dual-diagnosis motivational interviewing and integrated group therapy for jail inmates with co-occurring substance use and mental health disorders and to evaluate the feasibility of implementing the adapted interventions and associated research and communication protocols.

ELIGIBILITY:
Inclusion Criteria:

* (1) drug or alcohol abuse or dependence and SMI (major depressive disorder; depressive disorder not otherwise specified [NOS]; bipolar disorder I, II, or NOS; schizophrenia spectrum disorder; schizoaffective disorder; schizophreniform disorder; brief psychotic disorder; delusional disorder; or psychotic disorder NOS);
* (2) resident of Wake County and detained in The Jail;
* (3) >18 years of age; (4) able to speak/read English; and (5) able to provide informed consent.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability | Study months 21 through 34
  Client Satisfaction Questionnaire-8, Narrative Evaluation of Intervention Interview

SECONDARY OUTCOMES:
Feasibility of Adapted Interventions | Study months 21 through 34
  How successfully can the adapted interventions be implemented (Focus Group interviews)
Fidelity | Study months 21 through 34
  DDMI and IGT Adherence Forms
Substance use | Study months 20 through 30
  Addiction Severity Index
Psychiatric symptoms | Study months 20 through 30
  Brief Psychiatric Rating Scale
Health status | Study months 20 through 30
  SF-12
Service use | Study months 20 through 30
  Epidemiological Catchment Area Interview
Externalizing behaviors | Study months 20 through 30
  Triarchic Psychopathy Measure
Quality of life measure | Study months 20 through 30
  Heinrichs-Carpenter Quality of Life Scale, Plus
Arrest | Study months 20 through 30
  Self-report and official jail records
Treatment preferences | Study months 20 through 30
  Visual analog ranking of 8 different aspects of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Van Dorn, Ph.D., Principal Investigator — RTI International
Locations (1):
- RTI International, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Van Dorn RA, Desmarais SL, Rade CB, Burris EN, Cuddeback GS, Johnson KL, Tueller SJ, Comfort ML, Mueser KT. Jail-to-community treatment continuum for adults with co-occurring substance use and mental disorders: study protocol for a pilot randomized controlled trial. Trials. 2017 Aug 4;18(1):365. doi: 10.1186/s13063-017-2088-z. PMID 28778175